CLINICAL TRIAL: NCT03928093
Title: A Double-blind, Randomized, Cross-over, Feasibility Trial of Pregabalin for the Treatment of Recessive Dystrophic Epidermolysis Bullosa-associated Neuropathic Pain and Itch
Brief Title: Pregabalin Treatment for RDEB Pain and Itch
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Epidemolysis Bullosa Research Partnership (Other Government)
Responsible Party: Principal Investigator, Elena Pope, Dermatology section head, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000060628
Record Dates: First submitted 2019-03-27; First posted 2019-04-25 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Pain, Neuropathic; Itch; Epidermolysis Bullosa
MeSH Terms: conditions — Neuralgia; Pruritus; Epidermolysis Bullosa | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: there two treatment periods in the study. All of the study participants will receive pregabalin treatment during one of these two 10-week treatment periods, and placebo - during the other one.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigators, assessors and participants will be blinded to the intervention. The randomization will be done by the research pharmacist. Unblinding before the study completion is allowed only in case of serious adverse events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pregabalin followed by placebo (Experimental): The study has a crossover design. Participants in this arm will receive pregabalin during the first study treatment period for ten weeks and placebo during their second ten-week treatment period . The dose will depend on the participant's weight and phase of treatment period. Each treatment period consists of 4 weeks of escalating dose until the desired maximum , 4 weeks of active treatment and 2 weeks of titrating down.
  Interventions: Drug: Pregabalin
- Placebo followed by Pregabalin (Experimental): Participants will receive placebo during the first treatment period of the study(10 weeks) followed by 10 weeks of pregabalin treatment . The dose will depend on the participant's weight and phase of the treatment period . Each treatment period consists of 3 phases: 4 weeks of escalating dose until the desired maximum, 4 weeks of active treatment and 2 weeks of titrating down.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin /placebo capsules will be taken by mouth and will be prescribed for the study participants in the doses, depending on their weight and treatment phase: Participant < 25 kg at baseline will start with 50 mg per day, increasing the dose by 50 mg each week until their maximum dose 200 mg per day; Participants who are greater than or equal to 25 kg at baseline will start with 100 mg per day, increasing their dose by 50 mg each week until their target dose 300 mg per day is achieved. The study medication will be taken twice per day.The dose will be weaned down every 1-2 days by 25 mg in the last two weeks of each treatment period.
  Other Names: Placebo

SUMMARY:
Recessive dystrophic epidermolysis bullosa (RDEB) patients' quality of life is severely affected by neuropathic pain and itch, which have recently been demonstrated to be secondary to skin small fiber neuropathy. To date, there is no evidence on what the best agent is to control these symptoms. Based on the anecdotal data and safety profile, the investigators believe that pregabalin is a therapeutic agent that will be effective and safe in this population. The investigators propose to conduct a blinded study, using pregabalin versus placebo in which each patient serves as its own control (cross-over design). This is a feasibility study that will provide preliminary data on efficacy and safety of pregabalin in RDEB patients with neuropathic pain and itch and gather much needed data (dosage, titration schedule, outcome measures, etc) to inform the design of a larger cohort, controlled, multicenter trial.

DETAILED DESCRIPTION:
Neuropathic pain and itch are significant symptoms that affect RDEB patients' quality of life. To date, there is no evidence on what the best agent is to control these symptoms.

Based on the anecdotal data and the safety profile, the investigator believes that pregabalin is a therapeutic agent that will be effective and safe in this population.

This is a pilot, randomized, double-blinded, cross-over trial of pregabalin vs placebo for the treatment of RDEB associated neuropathic pain and itch. The study will run for 24 weeks and will have 4 separate phases with 6 overall visits: 1. Observation/wash out period (2 weeks); 2. ARM-1, ½ of the patients will receive pregabalin(A) and ½ the placebo (B) (10 weeks); 3. Wash out period (2 weeks) and 4. ARM-2 (patients who received placebo will receive pregabalin and pregabalin will receive placebo (10 weeks).

Patients will be recruited during the regular clinic visits or invited to participate via a letter followed by 2 phone calls.

1. Screening/Wash out period #1 (Visit 0)to assess eligibility criteria and the background pain and itch level (2 weeks), as well as the effectiveness of patients' "standard pain/itch interventions". Throughout this phase and the rest of the study, patients will receive pain and itch medications, except those that interfere with the pregabalin (see exclusion criteria).

   * Investigators will assess the eligibility criteria, including having moderate to severe pain (>4/10), the evidence of neuropathy using a thermal roller device ROLLTEMP2, Sometic, and a screening tool for neuropathic pain, the DN4 questionnaire 15 (Appendix 2).
   * Investigators will collect basic demographic data, medication information and disease severity using iscorEB clinician portion, a valid outcome measure that evaluates the disease severity 16 and EBDASI 17 ( Data collection form: Baseline/Screening Form)
   * Patients will be asked to report on their disease severity using iscorEB patient portion (all ages) that includes pain and itch domains and QOLEB 18 for those over 18 years of age (validated only for the adult population).
   * Patients will be instructed how to collect daily assessments of pain and itching for 14 days before the next visit. For the overall pain intensity assessment, the investigators will use a 100mm VAS, where 0 is no pain and 10- the worst pain ever experienced. For itch assessments, the investigators will ask patients to score each day, before going to bed, the degree of itching experienced that day using a 100 mm horizontal VAS where 0 is no itch and 10 is the worst itch.19 The investigators chose the single item for its reliability, validity and responsiveness to change. These values will represent patient's baseline pain (AvePain-00) and itch (AveItch-00).
2. ARM1 intervention study period (Visits 1 & 2): ½ of the patients will receive the active intervention (Pregabalin) and ½ the placebo. This phase will be of 10 weeks duration and will consist of 4 weeks of escalating dose until the desired maximum, 4 weeks of active treatment and 2 weeks of titration down (see titration schedule in the Appendix 1)Patients will receive either active intervention (pregabalin) or placebo including instruction of how to administer them.

   Visit 1: (Week 2)
   * Investigator will collect the data on pain and itching from the 2 weeks wash-out and will determine the average pain and itching of approximately 14 days prior to the study visit 1(AvePain-00, AveItch-00)
   * Patients will be asked to report on their disease severity using iscorEB patient portion and QOLEB for those over 18 years of age.
   * A team member will call patient twice a week during the escalation phase to inquire about adverse events
   * Patients will be instructed to collect daily assessments of pain, and itch for 7 days before next visit (~from weeks 9-10).

   Visit 2: (Week 10)
   * Patients will be instructed to contact investigator if experiencing any adverse events.
   * Investigator will collect the data on pain and itching from approximately 7 days prior to visit 2 (~weeks 9-10) and will determine the average pain and itching (AvePain-02, AveItch-02)
   * Patients will be asked to report on their disease severity using iscorEB patient portion and QOLEB for those over 18 years of age.
   * Adverse events (see potential risks, DCF follow up, patient's diary)
   * Patients will be instructed to collect daily assessments of pain, and itch for 7 days before next visit (~from weeks 13-14)
3. Wash out period #2 (2 weeks) Visit 3 (Week 14)

   * Investigator will collect the data on pain and itching and will determine the average pain and itching of approximately 7 days prior to the study visit 3 (AvePain-03, AveItch-03)
   * Patients will be asked to report on their disease severity using iscorEB patient portion and QOLEB for those over 18 years of age.
   * Investigator will collect adverse events (see potential risks, DCF follow up, patient's diary)
   * Patients will be instructed to collect daily assessments of pain, and itch for 7 days before next visit (~from weeks 21-22)
   * All study procedures at visit 3 will be similar to visit 1.
4. ARM2 intervention study period (Visits 4 & 5 (Week 22 and 24): patients randomized to placebo will receive pregabalin and those on placebo will get the pregabalin conducted similarly as in ARM1

   * All study procedures at visit 4 will be similar to visit 2
   * The outcome measures will be similar, but will be recorded as (AvePain-04, AveItch-04)
   * Weaning will be similar to ARM1
   * End of the Study visit: Visit 5 (Week 24) The outcome measures will be similar, but will be recorded as AvePain-05, AveItch-05)

ELIGIBILITY:
Inclusion Criteria:

* Age: > 8 - 40 years (we selected this range due to lack of data in younger population and the difficulty in getting patient reported outcomes in younger patients)
* Diagnosis of RDEB (by a dermatologist and/or EB specialist and/or genetic confirmation)
* Evidence of neuropathy defined by: thermal sensory loss (determined by a thermal roller, ROLLTEMP2, Sometic, Sweden) 14 and > 4/10 score using a screening tool for neuropathic pain, the DN4 questionnaire 15
* Pain intensity of > 4/10 on a 0-10 VAS scale measured daily (reduced frequency is also acceptable) at night over 2 weeks
* Itch intensity of > 4/10 on a 0-10 VAS scale measures daily (reduced frequency is also acceptable) at night over 2 weeks
* Consent to follow with study procedures

Exclusion Criteria:

* Intolerance and/or allergy to Pregabalin or gabapentin
* Lactose intolerance (placebo capsules contain lactose)
* Pregabalin use within 2 weeks before study enrolment
* Ongoing treatment with gabapentin, amitriptyline, duloxetine, nortriptyline, other tricyclics or SNRIs
* Medical conditions that would be considered as contraindications for pregabalin treatment (ischemic heart disease, cardiac dysrhythmia, glaucoma, history of urinary retention)
* Pregnancy
* History of use of restrictive substances or alcohol abuse
* Allergy to gelatin

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Difference in the mean pain scores between pregabalin and placebo group: VAS | 12 weeks
  It will be measured as difference in the mean pain values pre- and post-intervention for each group using the Visual Analog Scale (VAS).It is a 10 cm line with anchor statements on the left (no pain) and on the right (worst pain ever). The patient is asked to mark their pain level on the line.The pain is scored using the VAS by measuring the distance in centimeters (0-10) from the "no pain" anchoring point.

SECONDARY OUTCOMES:
Proportion of patients on pregabalin achieving a ≥75% reduction in their mean pain intensity score across last 7 days of treatment compared to baseline/wash-out | 12 weeks
  Proportion of patients on pregabalin achieving a ≥75% reduction in their mean pain intensity score across last 7 days of treatment compared to baseline/wash-out
Proportion of patients on pregabalin achieving a ≥50% reduction in their mean pain intensity score across last 7 days of treatment compared to baseline/wash-out | 12 weeks
  Proportion of patients on pregabalin achieving a ≥50% reduction in their mean pain intensity score across last 7 days of treatment compared to baseline/wash-out
Difference in the average pain score assessed using VAS between first and second treatment periods (period effect) | 24 weeks
  Difference in the average pain score assessed using VAS, reported by the patient between first and second treatment periods. Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (0 -no pain) and on the right (10- worst pain ever). The patient is asked to mark their pain level on the line. The pain is scored using the VAS by measuring the distance in centimeters (0-10) from the "no pain" anchoring point.
Proportion of patients on pregabalin achieving a ≥75% reduction in their mean itch intensity score across last 7 days of treatment compared to baseline/wash-out | 24 weeks
  Proportion of patients on pregabalin achieving a ≥75% reduction in their mean itch intensity score across last 7 days of treatment compared to baseline/wash-out.The intensity of itch is measured using the Visual Analog Scale for itch(VAS).It is a 10 cm line with anchor statements on the left (no itching) and on the right (worst possible itching). The patient is asked to mark the intensity of itch on the line. The itch is scored using the VAS by measuring the distance in centimeters (0-10)from the "no itch" anchoring point.
Proportion of patients on pregabalin achieving a ≥50% reduction in their mean itch intensity score across last 7 days of treatment compared to baseline/wash-out | 12 weerks
  Proportion of patients on pregabalin achieving a ≥50% reduction in their mean itch intensity score across last 7 days of treatment compared to baseline/wash-out
Difference in the average itch score as assessed using VAS between the first and the second treatment periods (period effect). | 24 weeks
  Difference in the average itch score as assessed using VAS( reported by the patient) between the first and the second treatment periods (period effect). The intensity of itch is measured using the Visual Analog Scale for itch (VAS).It is a 10 cm line with anchor statements on the left (0- no itching) and on the right (10 -worst possible itching). The patient is asked to mark the intensity of itch on the line. The itch is scored using the VAS by measuring the distance in centimeters (0-10) from the "no itch" anchoring point.
Changes in the Quality of Life in Epidermolysis Bullosa Questionnaire score(QOLEB) for patients >18yrs in the intervention versus placebo | 24 weeks
  Changes in the QOLEB for patients >18yrs in the intervention versus placebo. QOLEB is a measurement tool containing 17questions.Each question has a score range from 0-3.Total score range is between 0 and 51.
  iscorEB is a measurement tool for evaluating the disease severity in EB patient.It evaluates the cutaneous,mucosal and other organ impact of EB and includes clinician and patient reported outcomes in a single instrument. Score ranges between 0-120 for both reported outcomes.
Changes in iscorEB (instrument for scoring clinical outcomes for research of EB), patient portion score in the intervention versus placebo | 24 weeks
  iscorEB is a measurement tool for evaluating the disease severity in EB patient. It evaluates the cutaneous, mucosal and other organ impact of EB and includes clinician and patient reported outcomes in a single instrument. Score ranges between 0-120 for both reported outcomes. Patient portion of this instrument contains 15 questions. Each question has a score range from 0-8.Total score range for iscorEB patient portion is between 0 and 120. Reduction in iscorEB scores indicates improvement. An increase in score indicates deterioration.

OTHER OUTCOMES:
Correlation between pain score (as measured by VAS), iscorEB patient portion score and QOLEB (for patients over 18 yrs) total scores. | 24 weeks
  Correlation between pain score, as measured by Visual Analog Scale (VAS), iscorEB (instrument for scoring clinical outcomes for research of EB)- patient portion score, and Quality of Life in Epidermolysis Bullosa Questionnaire (QOLEB) score (for patients over 18 years). Please see full description of the mentioned instruments above.
Correlation between pain score( as measured by VAS) and iscorEB clinician portion score and Epidermolysis Bullosa Disease Activity and Scarring Index(EBDASI) score. | 24 weeks
  Correlation between pain score(as measured by Visual Analog Scale), iscorEB (instrument for scoring clinical outcomes for research of EB)- clinician portion score and EBDASI total score.Total EBDASI score ranges of 0-42, 43-106 and 107-506 corresponded to mild, moderate and severe disease respectively. Reduction in EBDASI activity scores of greater than 9 indicated clinically significant improvement. An increase of 3 in the activity score indicated deterioration. iscorEB is a measurement tool for evaluating the disease severity in EB patient. It evaluates the cutaneous, mucosal and other organ impact of EB and includes clinician and patient reported outcomes in a single instrument. Clinician score ranges between 0-120 between. Reduction in iscorEB scores indicates improvement. An increase in score indicates deterioration.
Proportion of patients experiencing adverse events, minor, severe and serious (life-threatening) | 24 weeks
  Proportion of patients experiencing adverse events
Proportion of patients that dropped out of the study as a result of an adverse event | 24 weeks
  Proportion of patients that dropped out of the study as a result of an adverse event
Correlation between itch score (as measured by VAS),iscorEB patient portion and QOLEB (for patients over 18 yrs) total scores. | 24 weeks
  Correlation between itch score( as measured by VAS),iscorEB patient portion, and QOLEB (for patients over 18 yrs.) total scores.
Correlation between itch score( as measured by VAS) and iscorEB clinician and Epidermolysis Bullosa Disease Activity and Scarring Index(EBDASI) | 24 weeks
  Correlation between itch score(as measured by VAS) and iscorEB clinician and EBDASI total scores. Total EBDASI score ranges of 0-42, 43-106 and 107-506 corresponded to mild, moderate and severe disease respectively. Reduction in EBDASI activity scores of greater than 9 indicated clinically significant improvement. An increase of 3 in the activity score indicated deterioration.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Calvo M, Tejos-Bravo M, Passi-Solar A, Espinoza F, Fuentes I, Lara-Corrales I, Pope E. Pregabalin for Neuropathic Pain and Itch in Recessive Dystrophic Epidermolysis Bullosa: A Randomized Crossover Trial. JAMA Dermatol. 2024 Dec 1;160(12):1314-1319. doi: 10.1001/jamadermatol.2024.3767. PMID 39441591